CLINICAL TRIAL: NCT03688997
Title: Expert Surgeons Versus Novice Residents: Validating a Novel Knot Tying Simulator for Vessel Ligation
Brief Title: Knot Tying Surgical Simulator for Vessel Ligation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Imri Amiel, Principal Investigator, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2646-15-SMC
Record Dates: First submitted 2018-09-21; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Surgery
Keywords: simulator; knot tying; vessel ligation; surgical training

STUDY DESIGN:
Intervention Model Description: Fifteen attending surgeons and 30 first year surgical residents were recruited to the study held at tertiary medical center during the years 2016-2017. The participants tied eight knots in different settings (Superficial vs. Deep) and techniques (One hand vs. two hands).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experts (Experimental): For the novice group, the investigators recruited 30 residents within their first year of surgical residency (Post-Graduate Year [PGY]-1) in general surgery, vascular surgery, plastic surgery, orthopedic surgery, cardio-thoracic surgery, gynecology and urology.
  The intervention administered was the use of a simulator by the participants.
  Interventions: Other: Simulator training
- Novice (Experimental): The expert's group included 15 attending surgical faculty members in the general surgery, vascular surgery, cardio-thoracic surgery and gynecology services.
  The intervention administered was the use of a simulator by the participants.
  Interventions: Other: Simulator training

INTERVENTIONS:
Other: Simulator training — bench-top simulator with computer acquired assessments, designed to allow novices to acquire basic surgical skills in knot tying. The simulator measures the forces used and applied on the tissue while ligating a vessel. Simulator training was included in both arms (expert and novice groups).

SUMMARY:
The investigators developed a bench-top knot tying simulator (KNOTI), with computer acquired assessment. Fifteen attending surgeons and 30 first year surgical residents were recruited to the study held at tertiary medical center during the years 2017-2018. The participants tied eight knots in different settings (Superficial vs. Deep) and techniques (One hand vs. two hands).

DETAILED DESCRIPTION:
The simulator is a bench-top simulator with computer acquired assessments, designed to allow novices to acquire basic surgical skills in knot tying. The simulator measures the forces used and applied on the tissue while ligating a vessel.

Each participant received instructions for approximately 10 minutes with a standardized and detailed explanation of the knot-tying technique. All knots were square knots (double-throw knot) using the same type of sutures (SOLFSILK 3.0). Participants were asked to tie two knots in four types: A superficial one hand square knot; A superficial two hand square knot; A deep one hand square knot; A deep two hand square knot.

For each knot six parameters were extracted from the sensor data: maximum upward force, maximum downward force, total upward force, total downward force, absolute non-zero force and performance time. Maximum force is the highest force applied during the knot tying.

Participants were not aware of what exact parameters the simulator was assessing. Novices were explained to avoid tissue rupture or loose knots. Knot integrity was evaluated by an investigator present during the simulation that discarded "air knots". Videos were reviewed by an investigator at post-study analysis to verify the appropriate technique and knot integrity.

ELIGIBILITY:
Inclusion Criteria:

* residents within their first year of surgical residency
* attending physicians from general surgery, vascular surgery, cardio-thoracic surgery and gynecology services.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Less extent of force while knot tying for vessel ligation | Through study completion, an average of one year.
  The simulator will measure the vertical forces (in Newton) exerted while tying 8 knots for vessel ligation.

SECONDARY OUTCOMES:
Identify peak force while knot tying for vessel ligation | Through study completion, an average of one year.
  The simulator will measure the maximum upward force (in Newton) used while tying 8 knots for vessel ligation.

CONTACTS AND LOCATIONS:
Overall Officials: Imri Amiel, MD, Principal Investigator — Sheba Medical Center

IPD SHARING:
Plan to Share IPD: No